CLINICAL TRIAL: NCT06007768
Title: Autoimmune and Inflammatory Response Biomarkers in Fabry Disease
Acronym: Bio-FAIR
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor
Other Study IDs: 284/21
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Immune response; Biomarkers; Quality of life; Inflammation
MeSH Terms: conditions — Fabry Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma (EDTA and lithium heparin) and peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fabry Disease: Patients with Fabry disease, older than 18 years, and without autoimmune or autoinflammatory diseases.
- Control: Subjects without Fabry disease or autoimmune/autoinflammatory diseases, matched for age (± 5 years) and sex.

SUMMARY:
The goal of this observational study is to understand the immune response in Fabry disease (FD). We want to find out how the immune response is related to the severity of FD and how it affects patients' quality of life and pain.

Main Questions the Study Aims to Answer:

* How are immune response markers linked to the health of FD patients?
* How is the immune response different between FD patients and healthy individuals?

Participants:

We will include 20 patients who have FD and are older than 18, and do not have other autoimmune or autoinflammatory diseases. We'll also include a comparison group of the same size who don't have FD, but are similar in age and sex to the FD group.

Participants with Fabry disease will be asked about their medical history and complete questionnaires. We will measure their vital signs and collect blood samples to study immune response markers. We'll also look at specific biomarkers related to FD.

Healthy participants will do similar tasks for comparison.

Comparison: Researchers will compare the immune response markers and other measurements between FD patients and healthy individuals to understand the differences and similarities.

Duration: The study will take place over 18 months to gather comprehensive information.

DETAILED DESCRIPTION:
Rationale: The immune response could play a relevant role in the pathophysiological mechanisms of Fabry disease (FD), although the relationship between the activated immune pathways and the clinical expression of the disease needs to be clarified. Knowledge of the immune response in FD could help to better understand the progression of the disease, identifying new biomarkers potentially useful in the clinical follow-up of these patients.

Study design: Observational cross-sectional study with a control group. Study subjects: Target group: patients with Fabry disease, older than 18 years and without autoimmune or autoinflammatory diseases. Control group: subjects without Fabry disease matched for age (± 5 years) and sex.

Sample size: n=40 (20 patients with Fabry disease + 20 controls).

Objectives:

1. To study the relationship between immune response biomarkers and the clinical status of the patient, as measured by the MSSI scale (Mainz Severity Score Index) or by markers of target organ damage (clinical, biochemical and imaging parameters).
2. To characterize the immune response profile by circulating biomarkers of subjects with Fabry disease (FD) compared to healthy subjects.
3. To compare circulating biomarker values with those measured in PBMC (Peripheral Blood Mononuclear Cells) culture supernatant from patients with FD.
4. To evaluate the relationship between biomarkers of the immune response and the concentration of specific Fabry disease markers (Lyso-Gb3).
5. To evaluate the association between immune response biomarkers and quality of life and neuropathic pain in FD patients.

Variables: Demographics, vital signs, anthropometric data, FD medical history, questionnaires, clinical biochemical variables, biochemical markers of autoimmunity, specific markers of FD (Lyso-Gb3), immune response markers and markers of target organ damage.

Duration: 18 months

ELIGIBILITY:
For the Fabry Disease (FD) group:

Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of Fabry disease (enzymatic or genetic).
* Having signed the informed consent, after having received all the information concerning the study.

Exclusion Criteria:

* Autoimmune or autoinflammatory disease or patients with transplanted organs (corneal transplant excluded) and under additional immunosuppressive treatment.
* Acute cardiovascular event or major surgery in the 90 days prior to inclusion in the study.
* Serious intercurrent diseases such as HIV, COVID-19, cancer under active treatment, severe anemia, severe hepatic, respiratory or renal failure, or other pathologies that, at the investigator's discretion, could interfere with the objectives of the study.

For the Control group:

• Participants must not meet any of the exclusion criteria applied to the target (FD) population and must sign, prior to inclusion, the informed consent form after having received all the information concerning the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of consecutive patients with Fabry Disease (FD) under follow-up in the Internal Medicine Department of the Hospital Universitario Ramon y Cajal.
  In addition, a Control group of subjects without Fabry disease will be included, among those who come to donate blood at the Hospital Universitario Ramón y Cajal.
  Controls will be matched for age (± 5 years) and sex with FD patients.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
High-sensitivity C-reactive protein (hsCRP) | Day 1 (one cross-sectional examination only)
  High-sensitivity C-reactive protein (hsCRP), measured in mg/L.
Tumor necrosis factor (TNF) | Day 1 (one cross-sectional examination only)
  Tumor necrosis factor (TNF), measured in pg/mL.
Interleukin 6 (IL-6) | Day 1 (one cross-sectional examination only)
  Interleukin 6 (IL-6), measured in pg/mL.
Interferon gamma (IFN-γ) | Day 1 (one cross-sectional examination only)
  Interferon gamma (IFN-γ), measured in pg/mL.
Vascular cell adhesion protein 1 (VCAM-1) | Day 1 (one cross-sectional examination only)
  Vascular cell adhesion protein 1 (VCAM-1), measured in ng/mL.

SECONDARY OUTCOMES:
Globotriaosylsphingosine (Lyso-Gb3) | Day 1 (one cross-sectional examination only)
  The globotriaosylsphingosine (Lyso-Gb3), the deacylated derivative of Gb3, measured in plasma (ng/mL).
Brain natriuretic peptide (BNP) | Day 1 (one cross-sectional examination only)
  Brain natriuretic peptide (BNP), measured in pg/mL.
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | Day 1 (one cross-sectional examination only)
  N-terminal prohormone of brain natriuretic peptide (NT-proBNP), measured in pg/mL.
Cystatin C | Day 1 (one cross-sectional examination only)
  Cystatin C, measured in mg/dL.
EuroQol Health-Related Quality of Life (EQ-5D-5L) | Day 1 (one cross-sectional examination only)
  EQ-5D-5L is a standardised measure of health-related quality of life. The EQ-5D-5L essentially consists of a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, and five levels in these dimensions, and EQ-5D visual analogue scale (EQ VAS).
  A numerical value will be derived for each EQ-5D-5L health state (ranges from 1 representing full health to 0 representing dead) to reflect how good or bad a health state is according to the preferences of the general population in Spain.
  EQ VAS ranges from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
11-point numerical rating scale (NRS-11) score of neuropathic pain | Day 1 (one cross-sectional examination only)
  The Numeric Pain Rating Scale is a unidimensional measure of pain intensity in adults. The 11-point numerical rating scale (NRS-11) scores neuropathic pain ranging from '0' representing "no pain" to '10' representing "pain as bad as you can imagine".
Mainz Severity Score Index (MSSI) | Day 1 (one cross-sectional examination only)
  The Mainz Severity Score Index (MSSI) is an instrument for quantifying the overall severity of the signs and symptoms of Fabry disease. The MSSI assigns scores based on the presence and severity of signs and symptoms in four areas: general, neurologic, cardiovascular, and renal. Each of the signs and symptoms is weighted in accordance with its relationship to morbidity.
  MSSI scoring ranges from 0 (healthy) to 76 (maximum severity), and it is divided into severity bands of mild (<20), moderate (20-40), and severe (>40) affliction.

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Lopez Rodriguez, MD PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available for sharing upon reasonable request at the discretion of the Principal Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available one year after publication of the main results, during 5 years.
Access Criteria: Data will be available for sharing with investigators seeking to verify analyses or to conduct additional analyses that are appropriate to the nature of these data. Data will be made available for sharing upon request.

REFERENCES:
- [Background] Rozenfeld P, Feriozzi S. Contribution of inflammatory pathways to Fabry disease pathogenesis. Mol Genet Metab. 2017 Nov;122(3):19-27. doi: 10.1016/j.ymgme.2017.09.004. Epub 2017 Sep 13. PMID 28947349
- [Background] De Francesco PN, Mucci JM, Ceci R, Fossati CA, Rozenfeld PA. Fabry disease peripheral blood immune cells release inflammatory cytokines: role of globotriaosylceramide. Mol Genet Metab. 2013 May;109(1):93-9. doi: 10.1016/j.ymgme.2013.02.003. Epub 2013 Feb 13. PMID 23452955
- [Background] Mauhin W, Lidove O, Masat E, Mingozzi F, Mariampillai K, Ziza JM, Benveniste O. Innate and Adaptive Immune Response in Fabry Disease. JIMD Rep. 2015;22:1-10. doi: 10.1007/8904_2014_371. Epub 2015 Feb 18. PMID 25690728
- [Background] Ge W, Li D, Gao Y, Cao X. The Roles of Lysosomes in Inflammation and Autoimmune Diseases. Int Rev Immunol. 2015;34(5):415-31. doi: 10.3109/08830185.2014.936587. Epub 2014 Jul 30. PMID 25075736
- [Background] Simonetta I, Tuttolomondo A, Daidone M, Pinto A. Biomarkers in Anderson-Fabry Disease. Int J Mol Sci. 2020 Oct 29;21(21):8080. doi: 10.3390/ijms21218080. PMID 33138098
- [Background] Loso J, Lund N, Avanesov M, Muschol N, Lezius S, Cordts K, Schwedhelm E, Patten M. Serum Biomarkers of Endothelial Dysfunction in Fabry Associated Cardiomyopathy. Front Cardiovasc Med. 2018 Aug 15;5:108. doi: 10.3389/fcvm.2018.00108. eCollection 2018. PMID 30159316
- [Background] Shen JS, Meng XL, Moore DF, Quirk JM, Shayman JA, Schiffmann R, Kaneski CR. Globotriaosylceramide induces oxidative stress and up-regulates cell adhesion molecule expression in Fabry disease endothelial cells. Mol Genet Metab. 2008 Nov;95(3):163-8. doi: 10.1016/j.ymgme.2008.06.016. Epub 2008 Aug 15. PMID 18707907
- [Background] Weidemann F, Beer M, Kralewski M, Siwy J, Kampmann C. Early detection of organ involvement in Fabry disease by biomarker assessment in conjunction with LGE cardiac MRI: results from the SOPHIA study. Mol Genet Metab. 2019 Feb;126(2):169-182. doi: 10.1016/j.ymgme.2018.11.005. Epub 2018 Nov 12. PMID 30594474
- [Background] Chimenti C, Scopelliti F, Vulpis E, Tafani M, Villanova L, Verardo R, De Paulis R, Russo MA, Frustaci A. Increased oxidative stress contributes to cardiomyocyte dysfunction and death in patients with Fabry disease cardiomyopathy. Hum Pathol. 2015 Nov;46(11):1760-8. doi: 10.1016/j.humpath.2015.07.017. Epub 2015 Aug 4. PMID 26362204
- [Background] Yogasundaram H, Nikhanj A, Putko BN, Boutin M, Jain-Ghai S, Khan A, Auray-Blais C, West ML, Oudit GY. Elevated Inflammatory Plasma Biomarkers in Patients With Fabry Disease: A Critical Link to Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2018 Nov 6;7(21):e009098. doi: 10.1161/JAHA.118.009098. PMID 30571380
- [Background] Chen KH, Chien Y, Wang KL, Leu HB, Hsiao CY, Lai YH, Wang CY, Chang YL, Lin SJ, Niu DM, Chiou SH, Yu WC. Evaluation of Proinflammatory Prognostic Biomarkers for Fabry Cardiomyopathy With Enzyme Replacement Therapy. Can J Cardiol. 2016 Oct;32(10):1221.e1-1221.e9. doi: 10.1016/j.cjca.2015.10.033. Epub 2015 Nov 10. PMID 26919792